CLINICAL TRIAL: NCT04342793
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase 2a Study to Explore the Safety and Efficacy of ALS-L1023 in Patients With Non-alcoholic Steatohepatitis (NASH)
Brief Title: A Study to Evaluate the Efficacy and Safety of ALS-L1023 in Subjects With NASH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AngioLab, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AL101-NASH
Record Dates: First submitted 2020-04-06; First posted 2020-04-13 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — ALS-L1023

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo oral tablet
- ALS-L1023 1,200mg (Experimental): ALS-L1023 600mg twice a day
  Interventions: Drug: ALS-L1023 1,200mg
- ALS-L1023 1,800mg (Experimental): ALS-L1023 900mg twice a day
  Interventions: Drug: ALS-L1023 1,800mg

INTERVENTIONS:
Drug: Placebo oral tablet — Placebo
  Other Names: Placebo
  Arms: Placebo
Drug: ALS-L1023 1,200mg — ALS-L1023
  Other Names: ALS-L1023 tablet
  Arms: ALS-L1023 1,200mg
Drug: ALS-L1023 1,800mg — ALS-L1023
  Other Names: ALS-L1023 tablet
  Arms: ALS-L1023 1,800mg

SUMMARY:
The main objective of this study is to evaluate safety and efficacy of ALS-L1023 in patients with Non-alcoholic steatohepatitis

DETAILED DESCRIPTION:
Besides the main objectives, there are other objectives as follows:

1. To evaluate efficacy of ALS-L1023 for liver fibrosis and steatosis by noninvasive imaging biomarker MRI-PDFF and MRE
2. To determine optimized dose of ALS-L1023 in NASH disease

ELIGIBILITY:
Inclusion Criteria:

* Men or women ages 19 and over, under 75 years of age
* Patients diagnosed with NAFLD on abdominal ultrasonography and MRI
* Patients show presence of hepatic fat fraction as defined by ≥ 8% on MRI-PDFF and liver stiffness as defined by ≥ 2.5 kPa on MRE at Screening

Exclusion Criteria:

* Any subject with current, significant alcohol consumption or a history of significant alcohol consumption for a period of more than 3 consecutive months any time within 2 year prior to screening will be excluded
* Chronic liver disease (including hemochromatosis, liver cancer, autoimmune liver disease, viral hepatitis A, B, alcoholic liver disease
* Uncontrolled diabetes mellitus as defined by a HbA1c ≥ 9.0％ at Screening
* Patients who are allergic or hypersensitive to the drug or its constituents
* Pregnant or lactating women

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Change in liver fat percentage measured by MRI-PDFF | baseline, 24 weeks
  Liver fat is measured by MRI-PDFF
Change in liver fibrosis measured by MRE | baseline, 24 weeks
  Liver fibrosis is measured by Magnetic Resonance Enterography
Change in visceral fat area measured by MRI | baseline, 24weeks
  Visceral fat area is measured by MRI
Changes in serum concentrations of ALT and AST | baseline, 24weeks
  ALT and AST concentrations in serum are measured

SECONDARY OUTCOMES:
Change in serum concentration of Pro-C3 | baseline, 24weeks
  Pro-C3 concentration in serum is measured
Change in serum concentration of CK-18 | baseline, 24weeks
  CK-18 concentration in serum is measured
Change in insulin sensitivity determined by HOMA-IR | baseline, 24weeks
  Insulin sensitivity is determined by Homeostatic Model Assessment for Insulin Resistance
Change in serum concentration of Leptin | baseline, 24weeks
  Concentration of Leptin in serum is measured
Changes in serum concentrations of ALT and AST | baseline, 8weeks, 16weeks
  ALT and AST concentrations in serum are measured
Changes in serum concentrations of TG and TC | baseline, 8weeks, 16weeks, 24weeks
  Triglyceride and Total Cholesterol concentrations in serum are measured
Change of NAFLD fibrosis score(NFS) | baseline, 8weeks, 16weeks, 24weeks
  NFS is measured
Change in serum concentration of Ghrelin | baseline, 24weeks
  Concentration of Ghrelin in serum is measured
Change in serum concentration of Adiponection | baseline, 24weeks
  Concentration of Adiponection in serum is measured

CONTACTS AND LOCATIONS:
Overall Officials: Dae Won Jun, Ph. D., Principal Investigator — Hanyang University
Locations (1):
- Hanyang University Seoul Hospital, Seoul, South Korea